CLINICAL TRIAL: NCT06502093
Title: Relationship Between Hospital Foodservice, Patient Satisfaction, and Malnutrition Risk: A Pilot Study in Hospital
Brief Title: Hospital Foodservice, Patient Satisfaction, and Malnutrition Risk
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Head of Nutrition and Dietetic Department, Clinical Assistant Professor, Istanbul Bilgi University
Other Study IDs: FOODSAT
Record Dates: First submitted 2024-07-03; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Food Services; Malnutrition
Keywords: Nutritional Assessment; Food Services; Malnutrition; Patient Satisfaction
MeSH Terms: conditions — Malnutrition; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study Group: * Aged 18-65,
  * Volunteers at the Isparta City Hospital
  * Patients who were hospitalized in neurology, internal medicine, general surgery, cardiovascular surgery, and chest disease clinics for at least seven days
  Interventions: Other: Observational Malnutrition Screening and Foodservice Satisfaction

INTERVENTIONS:
Other: Observational Malnutrition Screening and Foodservice Satisfaction — Patients asked Acute Care Hospital Foodservice Patient Satisfaction Questionnaire and malnutrition risk assessed with NRS-2002 screening tool.

SUMMARY:
Malnutrition is the body's inability to absorb necessary nutrients, often due to disease, hunger, aging, or other factors. The European Society for Clinical Nutrition and Metabolism (ESPEN) focuses on the malnutrition aspect [1,2]. Unidentified or unmonitored malnutrition before hospitalization, complications affecting eating, patient inability to eat regularly due to exams/treatments, delayed meal times, psychological factors, hospital stay duration, lack of nutrition awareness, prejudices against hospital meals, etc., can lead to hospital malnutrition. Patient-related issues and lack of dietitian referrals may contribute, with food service problems being a key factor in nutritional decline [3,4]. The critical factors affecting the patient's food appreciation include the appearance, presentation, taste, consistency, texture, and temperature. In cases where patient expectations and satisfaction are not met, a decrease in food consumption and an increase in the amount of leftovers are observed. It has been observed that if the organoleptic properties and presentation style of the food offered to the patient are good, the patients evaluate the food as high quality, and their satisfaction with the food increases [5]. As a result, not being able to consume food due to lack of meal satisfaction means that the energy and elements that the patient needs are not taken into the body, which increases the patient's risk of malnutrition [4]. Effective hospital meal provision is crucial in preventing malnutrition, as emphasized by ESPEN. One of the most essential duties of the dietitian is to supervise every stage of food services to ensure the consumption of foods suitable for medical nutrition treatment of the hospitalized patient [6,7].

This study aimed to determine the role and effect of hospital food services on inpatient malnutrition. For this purpose, NRS-2002 screening was performed on 310 inpatients within three days after admission. NRS-2002 is a comprehensive screening test that the ESPEN recommends for hospitalized patients. Along with the second NRS-2002 screening, a food service satisfaction survey was administered to patients. The results of both NRS-2002 screening and satisfaction surveys were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* volunteers patients
* Patients who were hospitalized for at least seven days

Exclusion Criteria:

* Patients with a hospital stay of less than seven days,
* receiving oral intake restrictive treatment,
* patients in the terminal phase,
* patients under 18 years of ages,
* patients over 65 years of ages.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized in neurology, internal medicine, general surgery, cardiovascular surgery, and chest disease clinics.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
NRS-2002 Screening Tool | NRS-2002 was administered for the first time 2 days after the patients were hospitalized. It was repeated for the second time 1 week later.
  NRS-2002 is a malnutrition assessment tool developed by Kondrup et al. As a result of the screening test, patients are classified as having no risk of malnutrition (<3 points) and having a risk of malnutrition (≥3 points)
Acute Care Hospital Foodservice Patient Satisfaction Questionnaire (ACHFPSQ) | The scale was administered once, 9 days after hospitalization, together with the NRS-2002 second screening.
  Acute Care Hospital Foodservice Patient Satisfaction Questionnaire (ACHFPSQ), developed by Capra et al. It is evaluated out of a total of 100 points. The increase in the patient's scale score in each sub-dimension means that satisfaction with hospital food services also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Demirel, PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon reasonable request from corresponding author.

REFERENCES:
- [Background] Kruizenga HM, Seidell JC, de Vet HC, Wierdsma NJ, van Bokhorst-de van der Schueren MA. Development and validation of a hospital screening tool for malnutrition: the short nutritional assessment questionnaire (SNAQ). Clin Nutr. 2005 Feb;24(1):75-82. doi: 10.1016/j.clnu.2004.07.015. PMID 15681104
- [Background] Klek S, Krznaric Z, Gundogdu RH, Chourdakis M, Kekstas G, Jakobson T, Paluszkiewicz P, Vranesic Bender D, Uyar M, Demirag K, Poulia KA, Klimasauskas A, Starkopf J, Galas A. Prevalence of malnutrition in various political, economic, and geographic settings. JPEN J Parenter Enteral Nutr. 2015 Feb;39(2):200-10. doi: 10.1177/0148607113505860. Epub 2013 Nov 4. PMID 24190900
- [Background] Sorensen J, Fletcher H, Macdonald B, Whittington-Carter L, Nasser R, Gramlich L. Canadian Hospital Food Service Practices to Prevent Malnutrition. Can J Diet Pract Res. 2021 Dec 1;82(4):167-175. doi: 10.3148/cjdpr-2021-013. Epub 2021 Jul 21. PMID 34286621
- [Background] Arends J, Baracos V, Bertz H, Bozzetti F, Calder PC, Deutz NEP, Erickson N, Laviano A, Lisanti MP, Lobo DN, McMillan DC, Muscaritoli M, Ockenga J, Pirlich M, Strasser F, de van der Schueren M, Van Gossum A, Vaupel P, Weimann A. ESPEN expert group recommendations for action against cancer-related malnutrition. Clin Nutr. 2017 Oct;36(5):1187-1196. doi: 10.1016/j.clnu.2017.06.017. Epub 2017 Jun 23. PMID 28689670
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Capra S, Wright O, Sardie M, Bauer J, Askew D. The acute hospital foodservice patient satisfaction questionnaire: the development of a valid and reliable tool to measure patient satisfaction with acute care hospital foodservices. Foodserv Res Int. 2005;16(1-2):1-14.